CLINICAL TRIAL: NCT00004474
Title: Phase III Randomized Study of Cyclophosphamide With or Without Antithymocyte Globulin Before Bone Marrow Transplantation in Patients With Aplastic Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Richard Champlin, University of Texas - MD Anderson Cancer Center
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 199/14004; RPCI-RP-9804; NCI-G98-1491; IBMTR-1
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2008-10

CONDITIONS: Aplastic Anemia
Keywords: Hematologic Disorders; Rare Disease
MeSH Terms: conditions — Anemia, Aplastic; Hematologic Diseases; Rare Diseases | interventions — Antilymphocyte Serum; Cyclophosphamide; Bone Marrow Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive cyclophosphamide IV over 60 minutes on Days -5 to -2 with antithymocyte globulin IV over 4 hours; then, after the last does cycophosphamide, participants will receive a bone marrow transplant over 60 to 120 minutes on Day 0.
  Interventions: Drug: Anti-thymocyte globulin; Drug: Cyclophosphamide; Procedure: Bone marrow transplantation
- 2 (Experimental): Participants will receive cyclophosphamide IV over 60 minutes on Days -5 to -2; then, after the last does cycophosphamide, participants will receive a bone marrow transplant over 60 to 120 minutes on Day 0.
  Interventions: Drug: Cyclophosphamide; Procedure: Bone marrow transplantation

INTERVENTIONS:
Drug: Anti-thymocyte globulin — Given via IV over 4 hours
  Arms: 1
Drug: Cyclophosphamide — Given via IV over 60 minutes on Days -5 to -2
Procedure: Bone marrow transplantation — Given on Day 0

SUMMARY:
OBJECTIVES:

I. Compare outcome, including graft failure, graft versus host disease, and survival of HLA-identical sibling bone marrow transplants for aplastic anemia using cyclophosphamide with or without antithymocyte globulin as a conditioning regimen.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, multicenter study. Patients are randomized to receive cyclophosphamide IV over 60 minutes on days -5 to -2 with or without antithymocyte globulin IV over 4 hours.

All patients then receive bone marrow over 60-120 minutes on day 0, 36 hours after the last dose of cyclophosphamide.

Patients are followed at day 100, at 6 months, and at 1 year posttransplant.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Severe aplastic anemia with the following criteria:

Hypocellular bone marrow with cellularity less than 20%

At least 2 of the following hematologic abnormalities:

* Neutrophil count no greater than 500/mm3
* Platelet count no greater than 20,000/mm3
* Reticulocyte count no greater than 50,000/mm3

HLA-identical sibling donor available

No clonal cytogenetic abnormalities, paroxysmal nocturnal hemoglobinuria, or myelodysplastic syndrome within 3 months of diagnosis of aplastic anemia

No congenital or constitutional aplastic anemia or Fanconi anemia

--Patient Characteristics--

Hepatic: Bilirubin less than 3 times upper limit of normal (ULN)

Renal: Creatinine less than 2 times ULN

Cardiovascular: Normal cardiac function

Other:

* No uncontrolled infection
* No severe concurrent disease
* HIV negative
* Fertile patients must use effective contraception

Max Age: 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 224
Dates: Start 1998-09; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Graft failure, graft versus host disease, and survival | Measured at Day 100, Month 6, and Year 1 post-transplant

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin